CLINICAL TRIAL: NCT06219109
Title: SeveriTy of Pulmonary Edema and Timing of Resolution in Patients With Severe Pre-eclampsia and Eclampsia (TIPER): A Physiological and Sonographic Prospective Observational Study
Brief Title: Pulmonary Edema Resolution in Severe Preeclampsia and Eclampsia
Acronym: TiPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Doctors with Africa - CUAMM (Other)
Responsible Party: Sponsor
Other Study IDs: Cuamm_02/23
Record Dates: First submitted 2023-09-08; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Eclampsia; Severe Pre-eclampsia
Keywords: Eclampsia; Preeclampsia; Lung ultrasound scan; Pulmonary oedema; Respiratory distress
MeSH Terms: conditions — Eclampsia; Pre-Eclampsia; Pulmonary Edema; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with severe preeclampsia or eclampsia suffer from pulmonary complications. Accurate assessment of patients with pulmonary involvement using lung ultrasound (LUS) and echocardiography could lead to earlier detection of pre eclampsia and eclampsia associated pulmonary oedema, ARDS (acute respiratory distress syndrome) and other pulmonary complications. here is currently limited evidence regarding the features, severity, aetiology and history of pulmonary oedema in this group of patients Data from this prospective observational study will facilitate the early recognition of pre-eclamptic and eclamptic patients with pulmonary involvement to implement optimal triage and early therapeutic choices in a limited resource setting (diuretics, escalation to non invasive or invasive ventilation, referral to HDU (High dependency unit) or ICU, dialysis) and potentially reduce unfavorable outcomes.

DETAILED DESCRIPTION:
Background - Maternal mortality from treatable causes concerning the critical care domain in low- income countries remains strikingly high. Maternal mortality in Sierra Leone is the highest in the world with 1,360 deaths per 100,000 born alive. The burden of obstetric-related critical care morbidity is also extremely high. In high-income countries less than 2% of intensive care unit admissions relate to obstetric illnesses, but these rise to 10% in resource-limited settings. Pre-eclampsia/eclampsia are hypertensive disorders of pregnancy, one of the 3 leading causes of maternal morbidity and mortality worldwide. Respiratory distress and pulmonary oedema are known complications of preeclampsia-eclampsia and their insurgence is a hallmark of severe disease. Pulmonary oedema is reported as a complication in 2.9% of patients with preeclampsia-eclampsia. Pulmonary involvement is associated with worse maternal and perinatal outcomes. Incidence is significantly higher in low income countries, rising to 12% due to poorer prenatal care and access to hospital care, and suboptimal diagnostic and management processes .

Aim - The primary aim is to describe the frequency of lung ultrasound consistent with pulmonary oedema and the timing of resolution after delivery.

Secondary aims include the assessment of the frequency of acute respiratory failure, other LUS findings beyond pulmonary edema, the assessment of oxygenation, the use of respiratory organ support strategies, assessment of cardiac function, and quantification of major direct/ indirect obstetric complications and of perinatal complications.

Hypothesis -

1. A high proportion (>20%) of patients show LUS signs consistent with pulmonary edema before delivery.
2. There is incomplete resolution of both clinical and ultrasound signs after in the 72 hours after delivery.

Setting - Princess Christian Maternity Hospital, Freetown, Sierra Leone Population - Female subjects, hospitalized with severe preeclampsia or eclampsia Methods - Single centre, prospective, cohort study of patients with severe pre-eclampsia and eclampsia. The expected duration of study is 1 year. All patients with suspected severe pre-eclampsia or eclampsia will undergo screening upon admission to HDU and the Eclamptic ward. Eligible patients will undergo a systematic clinical and LUS examination, straight after admission (before delivery). Clinical examination will focus on signs of respiratory, neurologic and cardiac failure. Lung ultrasound will be performed using a Butterfly ultrasound probe (Butterfly, USA). Lung ultrasound will be performed using the validated 12-region method. As heart failure is a common finding in preeclamptic women, echocardiography performed with a cardiac sector probe, will enable real-time assessment of maternal cardiac contractility and cardiac output. The same clinical, LUS and echocardiographic assessment will be repeated between 24 h to 72 h (after delivery). Whenever the pre-delivery timepoint is not feasible due to late arrival, emergency scenario or postpartum onset, the after delivery examination only will be performed.

ELIGIBILITY:
Inclusion Criteria:

- All patients with severe pre-eclampsia or eclampsia admitted to hospital Princess Christian Maternity Hospital

Exclusion Criteria:

* Patients with chronic hypertensive disorders
* Lung ultrasound not feasible, e.g., due to electricity breakdown, or absence of the trained sonographer or presence of subcutaneous emphysema,

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients hospitalized at PCMH with severe preclampsia and eclampsia will be enrolled if the applicable inclusion and exclusion criteria are met
Sampling Method: Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-02 (Estimated)

PRIMARY OUTCOMES:
Frequency of LUS consistent with pulmonary edema | during hospital stay, average of 1 month
  Frequency endpoint: proportion of patients with a LUS positive for pulmonary edema Severity: LUS aeration score
Timing of resolution after delivery | during hospital stay, average of 1 month
  Categorical: Fraction of patients with improvement or resolution of LUS findings.
  Numerical: delta LUS score between T1 and T2

SECONDARY OUTCOMES:
Frequency of acute respiratory failure in patients with Severe Pre eclampsia and in patients with Eclampsia | during hospital stay, average of 1 month
  Proportion of patients with acute respiratory failure
Frequency of other LUS findings | during hospital stay, average of 1 month
  Proportion of patients with
  * consolidations
  * isolated pleural effusion
  * minor LUS findings
Frequency of organ support strategies | during hospital stay, average of 1 month
  Fraction of patients that receive oxygen and/or CPAP (Continuous Positive Airway Pressure) and/or mechanical ventilation
Frequency of patients with abnormal cardiac function | during hospital stay, average of 1 month
  Defined as low cardiac index measured by ultrasound
Oxygenation assessment | during hospital stay, average of 1 month
  SpO2 (peripheral capillary oxygen saturation) to FiO2 (fraction of inspired oxygen) ratio
Frequency of Major Direct Obstetric Complications (MDOCs) | during hospital stay, average of 1 month
  Fraction of patients with at least one additional MDOC (antepartum hemorrhage, postpartum hemorrhage, sepsis, uterine rupture, obstructed labour)
Frequency of Indirect Obstetric complications | during hospital stay, average of 1 month
  Fraction of patients with at least one among stroke, severe malaria, acute kidney injury and cardiac insufficiency.
Frequency of perinatal complications | during hospital stay, average of 1 month
  Intra uterine fetal death (IUFD), Apgar score, Admission to special care baby unit (SCBU)

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Pisani, Principal Investigator — Doctors with Africa - CUAMM; Adeniji Adetunji Oladeni, Principal Investigator — University of Sierra Leone Teaching Hospitals Complex, Princess Christian Maternity Hospital
Locations (1):
- Princess Christian Maternity Hospital, Freetown, Sierra Leone

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-08): https://cdn.clinicaltrials.gov/large-docs/09/NCT06219109/Prot_SAP_000.pdf